CLINICAL TRIAL: NCT03702777
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 2a, Proof-of-Concept Study of ASP8302 in Subjects With Underactive Bladder
Brief Title: A Study of ASP8302 in Participants With Underactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8302-CL-0201; 2017-003693-13 (EudraCT Number)
Record Dates: First submitted 2018-10-05; First posted 2018-10-11 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Underactive Bladder
Keywords: Underactive Bladder; ASP8302
MeSH Terms: conditions — Urinary Bladder, Underactive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASP8302 100mg (Experimental): Participants will receive ASP8302 100mg capsules orally once daily for up to 4 weeks.
  Interventions: Drug: ASP8302
- Placebo (Placebo Comparator): Participants will receive ASP8302 matching placebo orally once daily for up to 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP8302 — Oral Capsule
  Arms: ASP8302 100mg
Drug: Placebo — Oral Capsule
  Arms: Placebo

SUMMARY:
The study objectives of this study are to evaluate the efficacy of ASP8302 compared with placebo in participants with underactive bladder (UAB), to investigate the safety and tolerability of ASP8302 compared with placebo in participants with UAB, to investigate the pharmacokinetics of ASP8302 in participants with UAB and to support the development of the UAB - Patient Reported Outcome (PRO).

DETAILED DESCRIPTION:
The study will comprise a screening visit, followed by a treatment period and a 2-week follow-up period, in total 8 weeks. Participants will visit the clinic at screening (visit 1) and every 2 weeks (visit 2, 3, 4, and 5). During the course of the study assessments will be performed at the visits.

ELIGIBILITY:
Inclusion Criteria:

At visit 1:

* Subject is diagnosed with UAB, defined as a bothersome chronic incomplete bladder emptying:

  * clinical condition is present for ≥ 6 months before screening, and
  * subject has a PVR ≥ 75 mL (measured by ultrasound after uroflowmetry; V1-PVRUS1).
* Subject on clean intermittent catheterization (CIC) should have been on CIC for at least 1 month and should be able to void spontaneously and not be completely dependent on CIC.
* Female subject must either:

  * Be of non-childbearing potential; post-menopausal (defined as at least 1 year without any menses for which there is no other obvious pathological or physiological cause) prior to screening, or documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy).
  * Or, if of childbearing potential; agrees not to try to become pregnant during the study and for 28 days after the final study drug administration, agrees to have a serum pregnancy test on all visits, have a negative serum pregnancy test at the screening visit, and agrees to consistently use 1 form of highly effective birth control starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* A sexually active male subject with female partner(s) of childbearing potential is eligible if he agrees to use a male condom starting at screening and continue throughout study treatment and for 90 days after the final study drug administration. If the male subject has not had a vasectomy or is not sterile, his female partner(s) is utilizing 1 form of highly effective birth control starting at screening and will continue throughout study treatment and for 90 days after the male subject receives the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration.
* Male subject with a pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 28 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in this study.

At visit 2:

* Subject has a PVR ≥ 100 mL (measured by catheterization, i.e., PVRC2).
* Subject has a VVST ≥ 50 mL and a bladder voiding efficiency ((BVE) (V2_BVE)) ≥ 10%. The VVST and V2_PVRC2 will be used to calculate V2_BVE = [VVST/(V2_PVRC2 + VVST)] times 100.

Exclusion Criteria:

At visit 1:

Related to lower urinary tract:

* Subject has significant BOO:

  * Subject has clinically significant urethral stricture (e.g., requiring surgery).
  * Female subject has uterus prolapse ≥ Grade 2 Shaw's system (up to or outside the introitus), moderate or severe cystocele (reaches or protrudes outside the introitus).
  * Male subject has a bladder outlet obstruction index (BOOI) ≥ 40 cm H2O on pressure flow study (PFS) (either performed on screening or within 12 months of the screening visit), or -if PFS is not available-a prostate volume (PV) of > 40 mL (Europe) > 30 mL (Japan) on ultrasound (either performed on screening or within 6 months of the screening visit). Note: if PFS is available and PV is above the cut-off level, the subject is not to be excluded if bladder outlet obstruction index (BOOI) is < 40.
  * Other condition that constitutes significant BOO.
* Subject is known to have urgency urinary incontinence that is clinically significant.
* Subject is known to have 1 or more bladder diverticuli that is/are clinically significant.
* Subject is known to have vesico-ureteral/renal reflux that is clinically significant.
* Subject has a urinary catheter in situ (including suprapubic catheters).
* Subject is known to have 1 of the following conditions as a primary cause for subject's UAB, or a condition that could potentially influence treatment outcome:

  * Neurological lesion or condition, including cerebrovascular accident, spinal lumbar disc hernia, spinal cord injury, multiple sclerosis, Parkinson's disease, Guillain-Barré syndrome, pudendal, hypogastric or pelvic nerve lesion. Diabetes mellitus is allowed if controlled with or without medical treatment (e.g., HbA1C < 7%).
  * Increased pelvic floor muscle activity during voiding (e.g., dyssynergic striated sphincteric activity/striated sphincteric activity during voiding, Fowler syndrome and pelvic floor muscle spasm).
  * Previous bladder surgery (e.g., bladder augmentation or reduction surgery, latissimus dorsi detrusor myoplasty). Prior Benign Prostatic Obstruction surgery or pelvic organ prolapse surgery is allowed if performed more than 6 months prior to screening.
  * Previous implant surgery for incontinence still in situ (e.g., tape, sling or artificial sphincter)
  * Significant active urological pain syndrome.
  * Previous pelvic radiation therapy.
* Dependence on use of a manual assistance method intended to improve bladder emptying (e.g., Credé's maneuver or suprapubic tapping).

Related to (previous or current) treatment and/or study drug:

* Subject is receiving 1 or more of the following non-medication therapies:

  * Electrostimulation therapy, e.g., neurostimulation/modulation or sacral nerve stimulation in the past 3 months.
  * Intravesical or injection based treatment (e.g., botulinum toxin injections in urethra or bladder in the past 12 months).
  * An ongoing bladder training program and/or pelvic floor muscle exercises, which started within 6 weeks prior to visit 1.
  * Muscle-derived stem cell injection in the bladder or urethra or bladder transplantation at any time prior to screening.
* Subject is using prohibited medications or subject is using restricted medications under conditions different to those specified in the concomitant medication section.
* Subject has a known or suspected hypersensitivity to ASP8302 or any of the inactive ingredients.

Related to concomitant conditions:

(Please note that these exclusion criteria do not require specific diagnostic evaluation during the screening visit, unless the subject presents with signs and symptoms suggesting the presence of this condition that were not present earlier.)

* Subject is known to have inflammatory bowel disease or clinically significant diarrhea.
* Subject is known to be immunocompromised due to conditions such as human immunodeficiency virus/acquired immune deficiency syndrome or hepatitis C.
* Subject has been diagnosed with clinically significant cardiovascular or cerebrovascular diseases within 6 months prior to visit 1, such as myocardial infarction, uncontrolled angina/coronary artery disease, significant ventricular arrhythmias and heart failure (New York Heart Association class III/IV).
* Subject has been diagnosed with clinically significant asthma, chronic bronchitis and/or chronic obstructive pulmonary disease.
* Subject is known to have a mean Fridericia corrected QT interval (QTcF) > 430 ms for males or > 450 ms for females, a pre-existing long QT syndrome or hypokalemia.
* Subject has a clinically significant abnormal 12-lead ECG.
* Subject has current or previous malignant disease of the pelvis. Subjects with a history of (non-pelvic) cancer are considered eligible if the subject has undergone therapy and the subject has been considered disease free for at least 5 years. Subject with completely excised basal cell carcinoma or squamous cell carcinoma of the skin and completely excised cervical cancer in situ are also considered eligible.
* Subject is known to have moderate to severe hepatic impairment (i.e., Child-Pugh class B or C).
* Subject is known to have severe renal impairment defined as estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m^2.
* Subject is known to have current or history of alcohol and/or drug abuse within the last 24 months prior to screening.
* Subject has clinical signs and symptoms of a urinary tract infection (UTI), which is combined with a result of urine test (e.g., positive urine culture containing > 100,000 cfu/mL in midstream urine). If a UTI is confirmed in the visit 1 sample, the run-in period should be stopped. After successful treatment of the UTI, the subject can be rescreened and if eligible enroll in the study. If the subject has asymptomatic bacteriuria (i.e., a positive urine culture without clinical signs and symptoms of a UTI), the subject should not be excluded.
* Subject has any of the following abnormal liver or kidney function parameters (as assessed in visit 1 sample):

  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or bilirubin increased to > 1.5 times the upper limit of normal (ULN).
  * Gamma glutamyltransferase (γ-GT) increased to > 3 times the ULN.
  * eGFR < 45 mL/min/1.73 m^2 based on the Modification of Diet in Renal Disease formula.

General:

* Subject has received investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject is known to have any condition, which makes the subject unsuitable for study participation.

At visit 2:

* Subject meets any of the exclusion criteria of visit 1.
* Subject has severe overactive bladder (OAB), i.e., experienced 3 or more episodes of urgency (Patient Perception of Intensity of Urgency Scale (PPIUS) grade 3 or 4), during the 3-day micturition diary period prior to visit 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in PVR After Standardized Bladder Filling Measured by Catheterization (PVRc2) at Week 4 | Baseline and week 4
  Volume of urine in the bladder after standardized bladder filling measured by catheterization (PVRc2).

SECONDARY OUTCOMES:
Voided Volume After Standardized Bladder Filling (VV_St) at Week 4 | Week 4
  VVst is thought to increase as the bladder emptying is improved. Standardizing the bladder filling is thought to increase accuracy in comparison with normal spontaneous bladder filling which will differ between time points. No multiplicity correction will be performed.
Bladder Voiding Efficiency Calculated With PVRc2 and VV-St (BVEc2) at Week 4 | Week 4
  Bladder voiding efficiency (BVE) is defined as the percentage of the total bladder capacity (BC) that is voided using the following formula: BVE = [volume voided (VV) / (PVR + VV)] x 100. BVEc2: BVE calculated for PVRc2 parameter i.e. BVEc2 = [VV_St / (PVRc2 + VV_St)] x 100.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (29):
- Germany (4):
  - Site DE49001, Duisburg
  - Site DE49002, Duisburg
  - Site DE49004, Gronau
  - Site DE49003, Mönchengladbach
- Japan (14):
  - Site JP81009, Nagoya, Aichi-ken
  - Site JP81008, Ōbu, Aichi-ken
  - Site JP81007, Yoshida-gun, Fukui
  - Site JP81006, Asahikawa, Hokkaido
  - Site JP81005, Sapporo, Hokkaido
  - Site JP81015, Sapporo, Hokkaido
  - Site JP81002, Kobe, Hyōgo
  - Site JP81012, Kurashiki, Okayama-ken
  - Site JP81011, Sayama, Osaka
  - Site JP81001, Shimotsuga-gun, Tochigi
  - Site JP81003, Fukuoka
  - Site JP81004, Kumamoto
  - Site JP81010, Saga
  - Site JP81013, Shizuoka
- Netherlands (3):
  - Site NL31003, Eindhoven
  - Site NL31002, Maastricht
  - Site NL31001, Rotterdam
- Poland (4):
  - Site PL48004, Mysłowice
  - Site PL48003, Piaseczno
  - Site PL48002, Szczecin
  - Site PL48001, Warsaw
- Slovakia (3):
  - Site SK42103, Košice
  - Site SK42101, Nitra
  - Site SK42102, Trenčín
- Site UK44002, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] van Till JWO, Arita E, Kuroishi K, Croy R, Oelke M, van Koeveringe GA, Chapple CR, Yamaguchi O, Abrams P. Muscarinic-3-receptor positive allosteric modulator ASP8302 in patients with underactive bladder. A randomized controlled trial. Neurourol Urodyn. 2022 Jun;41(5):1139-1148. doi: 10.1002/nau.24931. Epub 2022 Apr 14. PMID 35419807
- See also: Link to results on the Astellas Clinical Study Results Website. — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=400